CLINICAL TRIAL: NCT04806412
Title: The Prevalence of Oncodrivers in Malignant Pleural Effusions Associated With Non-small Cell Lung Cancer: A Prospective Study.
Brief Title: Oncodrivers in Malignant Pleural Effusions Associated With Non-small Cell Lung Cancer: A Prospective Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-889
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Malignant Pleural Effusion; Non-small Cell Lung Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Genes, fms

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized, cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: meassurement of PD-L1, ALK, EGFR — PD-L1 test will be performed on cell-blocks using PD-L1 antibodies 22C3 and staining platform Dako Omnis (Agilent, Glostrup -Denmark).
  ALK test will be performed on cell-blocks using staining platform Dako Omnis (Agilent, Glostrup- Denmark) and ALK antibodies "Origene" clone: OT1A4. Sample quality is assessed as for PD-L1.
  EGFR mutation analysis will be performed as follows: after tumor content evaluation of hematoxylin and eosin stained slides, relevant regions are macrodissected and subjected to a standard genomic DNA extraction procedure using the GeneRead DNA FFPE Kit (Qiagen). Samples will be analysed using the GeneRead QIAact Actionable Insights Tumor Panel (Qiagen)

SUMMARY:
Oncological treatment of patients with disseminated non-small cell lung cancer (NSCLC) is depending on the status of programmed death-ligand 1 (PD-L1), anaplastic lymphoma kinase (ALK) and epidermal growth factor receptor (EGFR), so called oncodrivers. These can be measured in pleural fluid, but the prevalence is uncertain. In a prospective study, the research team aim to measure PD-L1, ALK and EGFR in patients with pleural fluid cytology positive for NSCLC to report the prevalence. Also, the study will investigate if the chance of obtaining oncodriver status is depending on the volume analysed and how the lack of oncodrivers influence the following work-up.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, cohort study of patients with pleural effusion. Participants will be recruited from patients referred to the Pleura Clinic or admitted at the ward at the Department of Respiratory Medicine, Næstved Hospital, Næstved or at the Department of Respiratory Medicine, Zealand University Hospital, Roskilde, which is the two regional centres for workup of pleural effusions. Patients will be referred from either general practice or other hospital departments.

Pleural fluids with cytology positive for NSCLC will be tested for oncodrivers (for squamous cell carcinomas (SCC): PD-L1, for adenocarcinomas (AC): PD-L1, ALK and EGFR).

Follow-up will be 8 weeks after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pleural effusion known or suspected of association with NSCLC (pleural fluid cytology positive for cells from NSCLC)
* Patients must be able to give informed consent

Exclusion Criteria:

* Full oncodriver status measured in any pleural fluid in current work-up
* Inability to understand written or spoken Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-03-12 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of oncodriver status | assessed at 8 weeks follow-up
  Prevalence of oncodriver status (for squamous cell carcinomas (SCC): PD-L1, for adenocarcinomas (AC): PD-L1, ALK and EGFR) in pleural fluid in patients with cytology positive for pulmonary NSCLC

SECONDARY OUTCOMES:
Proportion of adequate and inadequate pleural fluid specimens | assessed at 8-week follow-up
Amounts of pleural fluid sent for analysis | assessed at 8-week follow-up
  Meassured in mL.
Correlation between amounts of pleural fluid sent to the pathologist and the chance of obtaining oncodriver status | assessed at 8-week follow-up
Number and type of additional diagnostic interventions including additional thoracentesis and cytological or histological biopsies | assessed at 8-week follow-up
Prevalence of oncodriver status in additional diagnostic interventions | assessed at 8-week follow-up
- Correlation between oncodriver status obtained in pleural fluid specimens and cytological or histological biopsies | assessed at 8-week follow-up
- Proportion of work-ups where the lack of obtained oncodriver status in pleural fluid specimens leads to additional diagnostic interventions including additional thoracentesis and cytological or histological biopsies | assessed at 8-week follow-up
- Proportion of work-ups where full oncodriver-status was obtained at the second thoracentesis | assessed at 8-week follow-up
- Proportion of patients with pleural fluid cytology negative of NSCLC, who is diagnosed with NSCLC. | assessed at 8-week follow-up
Patient assessed pain during thoracentesis | at day 1, 2 minutes after thoracentesis
  assessed by a questionnaire containing a VAS (Visual Analogue Scale, scale 0-10, 0 being no pain, 10 being the worse pain)
Proportion of patients experiencing pneumothorax | assessed at day 1, 10 minutes after thoracentesis and 8-week follow-up by evaluating the patient file
Proportion of patients experiencing bleeding | assessed at day 1, 10 minutes after thoracentesis and 8-week follow-up
Proportion of complications leading to admission | assessed at 8-week follow-up
  assessed by evaluating the patient file

CONTACTS AND LOCATIONS:
Locations (1):
- Næstved Sygehus, department of pulmonary medicine, Næstved, Region Sjælland, Denmark